CLINICAL TRIAL: NCT07043894
Title: A Prospective, Multicenter Study on the Efficacy and Safety of Romiplostim N01 for Chemotherapy-Induced Thrombocytopenia (CIT) in Children, Adolescents, and Young Adults (CAYA) With Hematological and Solid Tumors
Brief Title: Romiplostim N01 for Chemotherapy-Induced Thrombocytopenia in Pediatric Cancer Patients
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, SIDAN LI, Prof, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCH0011
Record Dates: First submitted 2025-06-21; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Solid Tumors; Hematological Tumor; Children; Adolescent; Chemotherapy Induced Thrombocytopenia
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Intervention Model Description: This study is a multicenter, open-label, single-arm trial. It plans to enroll 50 pediatric and adolescent patients with hematologic or solid tumors who are receiving high-intensity chemotherapy regimens. The study aims to evaluate the efficacy and safety of lusutrombopag N01 in treating chemotherapy-induced thrombocytopenia in this patient population. Patient data from all participating centers will be collected through an Electronic Data Capture (EDC) system. After signing the informed consent form, each subject will be assigned a unique screening number for identification throughout the study period.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Romiplostim N01 (Experimental): Participants receive weekly subcutaneous injections of romiplostim N01 (250 μg/vial; Qilu Pharmaceutical) starting at 2 μg/kg.
  Interventions: Drug: Romiplostim N01

INTERVENTIONS:
Drug: Romiplostim N01 — Participants receive weekly subcutaneous injections of romiplostim N01 (250 μg/vial; Qilu Pharmaceutical) starting at 2 μg/kg. Doses are adjusted weekly based on platelet counts: increased by 2 μg/kg if platelets are <50 × 10⁹/L, by 1 μg/kg if 50-99 × 10⁹/L, up to a maximum of 10 μg/kg. Treatment continues for up to 2 weeks but stops early if platelets reach ≥100 × 10⁹/L or increase by ≥30 × 10⁹/L from baseline.

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of romiplostim N01 in treating chemotherapy-induced thrombocytopenia (CIT) in children and adolescents/young adults (CAYA; aged 6-24 years) with hematologic malignancies or solid tumors. The main questions it aims to answer are:

* What proportion of participants achieve platelet count recovery (≥100×10⁹/L or an increase of ≥30×10⁹/L from baseline) within 3 weeks of romiplostim N01 treatment?
* What is the safety profile of romiplostim N01 in this population, including the incidence and severity of adverse events (especially bleeding and thrombosis)? This is a single-arm study (no comparison group). Researchers will assess the outcomes against predefined efficacy thresholds and historical data (e.g., a 60.7% response rate reported for another TPO-RA, hetrombopag).

Participants will:

* Receive weekly subcutaneous injections of romiplostim N01 (starting dose: 2 µg/kg).
* Have their romiplostim dose adjusted weekly based on platelet counts (increase by 1-2 µg/kg if platelets <99×10⁹/L, maximum dose 10 µg/kg, stop when target recovery is met).
* Undergo frequent monitoring, including blood tests (especially platelet counts), vital signs, physical exams, and assessment for adverse events and bleeding throughout the treatment and follow-up period.

DETAILED DESCRIPTION:
This prospective, multicenter, open-label, single-arm Phase II clinical trial investigates the efficacy and safety of romiplostim N01, a thrombopoietin receptor agonist (TPO-RA), for treating chemotherapy-induced thrombocytopenia (CIT) in children, adolescents, and young adults (CAYA) aged 6-24 years with hematologic malignancies or solid tumors. Romiplostim N01 binds to the c-MPL receptor on megakaryocytes and their precursors, activating JAK-STAT and MAPK-ERK signaling pathways to stimulate platelet production. Participants receive weekly subcutaneous injections of romiplostim N01 (250 μg/vial; Qilu Pharmaceutical) starting at 2 μg/kg. Doses are adjusted weekly based on platelet counts: increased by 2 μg/kg if platelets are <50 × 10⁹/L, by 1 μg/kg if 50-99 × 10⁹/L, up to a maximum of 10 μg/kg. Treatment continues for up to 2 weeks but stops early if platelets reach ≥100 × 10⁹/L or increase by ≥30 × 10⁹/L from baseline.

The study involves 10 site visits over 36 days, including screening (≤14 days), baseline (Day 0), treatment (Days 1, 3, 5, 8, 15), and follow-up (Days 22, 29, 36). Serial assessments include platelet counts (primary efficacy endpoint), hemoglobin, neutrophil levels, vital signs, physical examinations, ECOG performance status, and laboratory evaluations (renal/hepatic function, coagulation). Safety is rigorously monitored using NCI CTCAE v5.0 for adverse events (AEs), WHO bleeding scale for hemorrhage, and active surveillance for thrombosis. Rescue therapies (e.g., platelet transfusions, rhTPO, rhIL-11) are permitted per protocol-specified thresholds. Data are captured electronically (EDC system) with source verification per GCP standards.

Statistical analysis targets 50 participants (factoring in 10% attrition) to achieve 80% power (α=0.05, two-sided) for detecting superiority over historical controls (60.7% response rate for hetrombopag). The Full Analysis Set (FAS) includes all dosed participants, while the Per Protocol Set (PPS) excludes those with major deviations. The primary efficacy endpoint-proportion achieving platelet recovery (≥100 × 10⁹/L or Δ≥30 × 10⁹/L) by Week 3-is analyzed using Clopper-Pearson method for 95% CI, with missing data handled via non-responder imputation. Secondary analyses include time-to-recovery, nadir platelet values, transfusion requirements, and chemotherapy delays (descriptive statistics, Kaplan-Meier for time-to-event). Safety analyses focus on AE incidence, severity, and causality.

Conducted across 12 sites in China (e.g., Chinese Academy of Medical Sciences Cancer Hospital, Beijing Children's Hospital), the trial adheres to ICH-GCP, Declaration of Helsinki, and local regulations, with ethics committee approval and written informed consent. The operational timeline spans from first participant enrollment (July 2025) to study completion (September 2026). This study addresses a critical gap in CIT management for CAYA patients by prospectively evaluating romiplostim's dosing, efficacy, and safety profile in this population, with rigorous risk mitigation for thrombosis and bleeding events.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation with signed informed consent.
2. Aged 6-24 years, any gender.
3. ECOG performance status 0-2.
4. Histologically/cytologically confirmed non-myeloid malignancy requiring high-intensity chemotherapy with ≥1 myelosuppressive agent.
5. Patients with potential curative opportunity eligible for standard therapy.
6. Chemotherapy-induced thrombocytopenia (platelets <75×10⁹/L).
7. Anticipated survival ≥8 months.
8. Planned ≥2 additional chemotherapy cycles (21-/28-day cycles).
9. Laboratory parameters meeting:

   * Renal function: Cr ≤1.5×ULN; Ccr ≥55 mL/min.
   * Hepatic function:

     * Total bilirubin ≤1.5×ULN; ALT/AST ≤3×ULN;
     * For liver metastasis/cholangiocarcinoma: bilirubin ≤3×ULN, transaminases ≤5×ULN.
10. No participation in other drug trials within 4 weeks.
11. Good compliance with efficacy/safety follow-up per protocol.
12. Absence of severe complications (e.g., active GI bleeding/perforation, jaundice, obstruction, non-cancer fever >38°C).
13. Ability to comprehend and sign informed consent.

Exclusion Criteria:

1. Hematologic disorders (non-CIT etiology): AML, ITP, MDS, MPN, multiple myeloma, etc.
2. Non-CIT thrombocytopenia within 6 months (e.g., chronic liver disease, hypersplenism, infection, hemorrhage).
3. Known hypersensitivity to romiplostim N01 or excipients (cellulose-lactose, L-HPC, magnesium stearate, film coating).
4. Refractory cytopenias:

   * Hemoglobin <50 g/L despite RBC/EPO;
   * ANC <1.0×10⁹/L despite G-CSF.
5. Pelvic/spinal/large-field radiotherapy within 3 months.
6. Arterial/venous thrombosis within 3 months.
7. Severe cardiovascular disease (NYHA Class III-IV, arrhythmia with thromboembolic risk, post-CABG/stent) within 6 months.
8. Use of rhTPO, rhIL-11, or TPO-RAs (eltrombopag/avatrombopag/hetrombopag) within 2 weeks.
9. Investigator-assessed risks compromising safety/efficacy evaluation.

Ages: 6 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving platelet count recovery to ≥100×10⁹/L or an increase of ≥30×10⁹/L from baseline | 3 weeks

SECONDARY OUTCOMES:
Median time to platelets ≥100×10⁹/L or ≥30×10⁹/L increase from baseline | 3 weeks
Nadir platelet count | 3 weeks
Mean time to platelets ≥100×10⁹/L or ≥30×10⁹/L increase | 3 weeks
Platelet increase from baseline | 3 weeks
Median time to peak platelets | 3 weeks
Median time to nadir platelets | 3 weeks
Maximum platelet count | 3 weeks
Frequency of platelet transfusions | 3 weeks
Volume of platelet transfusions | 3 weeks
Proportion of patients with Cycle 2 delay ≥4 days due to thrombocytopenia | 6 weeks
Proportion of patients unable to start Cycle 2 due to thrombocytopenia | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sidan Li, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No